CLINICAL TRIAL: NCT05239208
Title: Effects of Oral Nutritional Supplementation With Dietary Counseling in 24-60 Months Old Children at Risk of Undernutrition
Brief Title: Effects of Oral Nutritional Supplementation in Children at Risk of Undernutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AL45
Record Dates: First submitted 2022-01-07; First posted 2022-02-14 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Undernutrition
MeSH Terms: conditions — Malnutrition | interventions — Population Groups; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Nutritional Supplement (ONS) Group (Experimental): Two servings per day in addition to dietary counseling
  Interventions: Other: Oral Nutrition Supplement (ONS) Group
- Control Group (Active Comparator): Dietary counseling
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Oral Nutrition Supplement (ONS) Group — Oral nutritional supplement specifically designed for nutritionally-at risk children and dietary counseling
  Arms: Oral Nutritional Supplement (ONS) Group
Other: Control Group — Dietary counseling
  Arms: Control Group

SUMMARY:
This prospective, randomized, controlled study will evaluate the effects of oral nutritional supplementation plus dietary counseling versus dietary counseling alone in children at nutritional risk.

ELIGIBILITY:
Inclusion Criteria:

* Children 24-60 months old
* Undernourished or at risk of undernutrition according to the WHO Growth Standards.
* Child's parent(s)/legal guardian (LG) is willing to abstain from giving additional non-study ONS other than the study product during the study intervention period.
* Child's parent(s)/LG is able and willing to follow study procedures and record data in parent diary and complete any forms or assessments needed throughout the study.
* Child's parent(s)/LG is not planning to relocate during the study period.
* Child's parent(s)/LG has voluntarily signed and dated an Informed Consent Form (ICF), approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) or other applicable privacy regulation authorization prior to any participation in the study.

Exclusion Criteria:

* Participant participates in another study that has not been approved as a concomitant study.
* Child is known to have galactosemia, be allergic or intolerant to any ingredient found in the study product.
* Child is currently drinking an Abbott product(s).
* Child had a history of preterm delivery, defined as a birth before 37 completed weeks of gestation as reported by parent(s)/LG.
* Child had birth weight < 2500 g or > 4000 g.
* Child whose either parent has BMI ≥ 27.5 kg/m2
* Child has continuous oral nutrition supplement (ONS) usage for at least 15 days in the past 1 month prior to screening. The standard ONS formula usually has an energy density of at least 1 kcal/mL, containing protein, carbohydrate and/or fat, as well as a wide range of micronutrients to supplement or use as the sole source of nutrition.
* Child has current acute or chronic infections including but not restricted to respiratory infections, diarrhea, acute and chronic Hepatitis B or C, HIV infection or tuberculosis.
* Child has been diagnosed with the following according to medical records or report by parent(s)/LG or the clinician's judgment:

  1. Severe gastrointestinal disorders such as celiac disease, short bowel syndrome, pancreatic insufficiency, or cystic (Exception: Intestinal parasites infection)
  2. Neoplastic, renal, hepatic or cardiovascular, hormonal or metabolic disorders, congenital disease or genetic disorders such as atrial or ventricular wall defects, Down's syndrome, or thalassemia
  3. Infantile anorexia nervosa, developmental disability, including physical disorders such as cerebral palsy, or developmental delay
  4. Disorders of hemoglobin structure, function or synthesis
  5. Clinically significant nutritional deficiency requiring specific treatment with another nutritional supplement (other than the study product) as diagnosed by the investigator.
  6. Any other clinically significant medical condition, which in the investigator's opinion, makes him or her unsuitable for inclusion in the study.

Ages: 24 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
Weight-for-Age Z-Score | Baseline to 120 Days
  Change in weight-for-age z-score

SECONDARY OUTCOMES:
Weight | Baseline to 240 Days
  Measured in Kg
Height | Baseline to 240 Days
  Measured in cm
Mid-Upper-Arm Circumference (MUAC) | Baseline to 240 Days
  Measured in cm
Weight-for-Height Measurement Calculations | Baseline to 240 Days
  Weight-for-height standard z-scores and percentiles
BMI-for-Age Measurement Calculations | Baseline to 240 Days
  BMI-for-age standard z-scores and percentiles
Height-for-Age Measurement Calculations | Baseline to 240 Days
  Height-for-age standard z-scores and percentiles
MUAMC Measurement Calculations | Baseline to 240 Days
  Mid-upper-arm-circumference-for-age standard z-scores and percentiles
Dietary Intake | Baseline to 240 Days
  Measured by 24-hour dietary recall
Appetite | Baseline to 240 Days
  Visual analog scale from Ate Very Little to Ate Very Much

OTHER OUTCOMES:
Body Composition | Baseline to 240 Days
  Measured by duel-energy x-ray absorptiometry
Bone Quality | Baseline to 240 Days
  Measured by duel-energy x-ray absorptiometry
Lower Leg Length | Baseline to 240 Days
  Measured in cm
Adverse Event Reporting | Baseline to 240 Days
  Parent reported adverse events
Healthcare Utilization | Baseline to 240 Days
  Number of sick days, healthcare visits, missed days school, missed days work
Physical Activity | Baseline to 240 Days
  Visual analog scale Not Active to Very Active
Child's Healthy Growth | Baseline to 240 Days
  Parent completed assessment of child's growth
Product Palatability | Study Day 1 to Study Day 240
  1, 5-point scale from Dislike it very much to Like to very much
Child's Sleep Assessment | Baseline to 240 Days
  Parent reported sleep habits
Early Childhood Behavior Questionnaire | Baseline to 240 Days
  6, 7-point Likert scale questions scored from Never to Always
Blood Biomarkers Amino Acid | Baseline to 240 Days
  Blood chemistry analysis of amino acid biomarkers
Blood Biomarkers Bone | Baseline to 240 Days
  Blood chemistry analysis of bone biomarkers
Hand Grip Strength | Baseline to 240 Days
  Measured in kg

CONTACTS AND LOCATIONS:
Overall Officials: Yen Ling Mandy Ow, PhD, Study Chair — Abbott
Locations (1):
- National Institute of Nutrition, Hà Nội, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ow MYL, Tran NT, Berde Y, Nguyen TS, Tran VK, Jablonka MJ, Baggs GE, Huynh DTT. Efficacy of long-term oral nutritional supplementation with dietary counseling on growth, body composition and bone mineralization in children with or at risk for undernutrition: a randomized controlled trial. Nutr J. 2025 Jul 14;24(1):110. doi: 10.1186/s12937-025-01133-5. PMID 40660276